CLINICAL TRIAL: NCT04908046
Title: Study Title A Multicenter, Open-label, Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of HMPL-295S1 in Treatment of the Patients With Advanced Malignant Solid Tumors
Brief Title: A Study of HMPL-295S1 in Patients With Advanced Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-295-00CH1
Record Dates: First submitted 2021-04-26; First posted 2021-06-01 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Advanced Malignant Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HMPL-295S1 open-label treatment arm (Experimental): During dose escalation, single-dose PK evaluation will be carried out firstly in each dose group.
  At the first therapeutic dose level, the single-dose treatment period is 5 days; from the 2nd dose level, the sponsor can determine the adjustment of single-dose treatment period to 3-5 days based on the available PK profile. Subsequently, the patients will receive oral HMPL-295S1 QD continuously in a therapeutic cycle of 28 days (Day 1 - 28 of each cycle), until reaching the criteria on the end of treatment. The patients in RP2D extended cohort will enter the consecutive treatment period directly.
  Interventions: Drug: HMPL-295S1 with dose escalation stage of 5mg up to 200mg, then expansion stage with recommended dose of therapeutic cycle of 28 days .

INTERVENTIONS:
Drug: HMPL-295S1 with dose escalation stage of 5mg up to 200mg, then expansion stage with recommended dose of therapeutic cycle of 28 days . — Patient starts the initial dose treatment with 5mg QD of HMPL-295S1, during dose escalation, single-dose PK evaluation will be carried out firstly in each dose group.
  At the first therapeutic dose level, the single-dose treatment period is 5 days; from the 2nd dose level, the sponsor can determine the adjustment of single-dose treatment period to 3-5 days based on the available PK profile.
  Subsequently, the patients will receive oral HMPL-295S1 QD continuously in a therapeutic cycle of 28 days (Day 1 - 28 of each cycle), until reaching the criteria on the end of treatment. The patients in RP2D extended cohort will enter the consecutive treatment period directly.

SUMMARY:
The objective of this study is to evaluate the safety, tolerability and PK profile of HMPL-295S1 and determine MTD and/or RP2D in patients with advanced malignant solid tumor. It will be extended to enroll 10-15 patients at this dose after RP2D is determined, as to further evaluate the safety of RP2D and the preliminary efficacy of HMPL-295S1. In addition, an exploratory study on the pharmacokinetic biomarkers of HMPL-295S1 is planned in this study.

DETAILED DESCRIPTION:
This study is expected to enroll 52-87 patients, including 30-60 patients for dose escalation, the enrollment will continue until about 12 patients in the dose group with response, as to determine RP2D (assuming the two dose groups will continue enrollment to 12 patients), additional 10-15 patients will be enrolled at the dose level of determined RP2D. The number of patients finally screened in the study will depend on the number of dose levels evaluated, occurrence of dose-limiting toxicity (DLT) in each dose group and the failure rate of screening.

ELIGIBILITY:
Inclusion Criteria:

All the following conditions must be met for enrollment:

1. Having understood this study adequately and being voluntary to sign the informed consent form;
2. Aged 18~75 years (inclusive);
3. Patients with histopathologically or cytologically confirmed advanced malignant solid tumors who have failure of standard of care or can not tolerate standard of care, or can not obtain standard of care for various reasons, or have no standard of care (regardless of previous surgery);
4. Having at least one measurable lesion (in accordance with the RECIST 1.1 criteria); note: the lesion previously irradiated can not be regarded as target lesion, unless unequivocal progression of disease is shown in radiological evidence after radiotherapy;
5. United States Eastern Cooperative Oncology Group (ECOG) Performance Status score ≤ 1;
6. Life expectancy ≥12 weeks based on investigator's judgment;
7. Having adequate bone marrow, hepatic and renal function (no transfusion of whole blood, blood components, blood products, no use of granulocyte colony-stimulating factor or other hematopoietic stimulator or drug for correction within two weeks prior to blood collection):

   * Absolute neutrophil count ≥1.5×109/L;
   * HGB≥90 g/L;
   * Platelet count ≥ 100×109/L;
   * Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN) [alanine aminotransferase (ALT) and aspartate aminotransferase (AST) need to be normal, serum total bilirubin needs to be ≤3 × ULN in the patients with Gilbert disease];
   * Serum ALT and/or AST ≤2.5 × ULN in the patients without hepatic metastasis (ALT and AST ≤5 ×ULN for those with liver metastasis);
   * Creatinine clearance ≥ 60 mL/min (calculated according to Cockcroft-Gault formula, see Appendix 11);
   * International normalized ratio (INR) ≤1.5, and activated partial thromboplastin time (aPTT) ≤ 1.5 ULN.
8. A man of childbearing potential and his heterosexual partner of childbearing age must agree to use effective contraceptive methods from the signature of informed consent form to 90 days after the last dose; any female of childbearing potential (including those who have received tubal ligation) must receive serum or urine pregnancy test and the result is negative within 7 days prior to the first dose of study drug; and she must agree to use effective contraceptive methods, for example, dual barrier contraceptive method, intrauterine device, etc., from the signature of informed consent form to 30 days after the last dose of study drug. Postmenopausal woman (age > 50 years and menopause for 1 year or above, in the absence of other biological or physiological reasons) and the woman receiving irreversible sterilization operation (including hysterectomy, bilateral ovariectomy or bilateral salpingectomy, but excluding tubal ligation) who is regarded as infertile, will not be restricted by this condition.

Exclusion Criteria:

* The patients can not participate in this study if any of the following conditions is met:

  1. Previous antitumor therapy meeting any of the following:

     1. Previous treatment with a ERK inhibitor and having PD;
     2. Receiving approved systematic antitumor therapy within 4 weeks prior to the first dose, including chemotherapy, targeted therapy, immunotherapy, biotherapy, etc. (elution for two weeks for hormone therapy or treatment with traditional Chinese medicine and Chinese patent drug with clear antitumor indication);
     3. In the treatment period of other interventional clinical study (including small molecular chemical drug and macromolecular antibody) within 4 weeks prior to the first dose. Patients can be enrolled in this study if they are involved in non-interventional clinical study (e.g., epidemiological study); and can also be enrolled if they stay in the survival follow-up period of one interventional clinical study.
     4. Having received major surgery or radical radiotherapy (except for the palliative radiotherapy for bone metastasis) within 4 weeks prior to the first dose.
  2. Toxicity associated with previous antitumor therapy (including surgery, chemotherapy, radiotherapy, targeted therapy and immunotherapy) not recovered to ≤ CTCAE grade 1, except for alopecia and peripheral neuropathy. The peripheral neurotoxicity needs to be recovered to ≤ CTCAE grade 2 in the patients who have been previously treated with platinum;
  3. Patients with central nervous system (CNS) malignant tumor or malignant solid tumor with known CNS metastasis;
  4. Combined with other malignant tumor or having a history of other malignant tumor within 2 years prior to study screening (not including the basal or squamous cell carcinoma of skin, non-melanoma skin cancer, papillary thyroid carcinoma that have been appropriately treated, or radically resected cervical carcinoma in situ and ductal carcinoma in situ);
  5. Known history of clinically significant liver disease, including viral or other hepatitis, except the following patients:

     * HBsAg positive patients can be enrolled if the polymerase chain reaction (PCR) test of hepatitis B virus (HBV) DNA is negative. The investigator can provide preventive or therapeutic antiviral therapy based on patient's condition and diagnostic routines during study treatment;
     * Patients with positive hepatitis C virus (HCV) antibody can be enrolled if the PCR test of HCV RNA is negative.
  6. Patients infected by human immunodeficiency virus (HIV);
  7. Presence of active bacterial, fungal or viral infection requiring systematic treatment within one week prior to the first dose;
  8. Use of CYP3A potent inducer within 2 week or 5 half-lives (whichever is longer, 3 weeks needed for St. John's wort) prior to the first dose, see (Appendix 5);
  9. Use of CYP3A, P-gp potent inhibitor or sensitive substrate of P-gp, BCRP, MATE 2-K, CYP3A, CYP2C8/OATP1B1 and CYP2D6/CYP3A within one week or three half-lives (whichever is longer) prior to the first dose, this exclusion criterion will be adjusted in accordance with the actual dose of HMPL-295S1 and determined plasma concentration during the clinical study (see Appendix 5);
  10. Meeting any of the following criteria for cardiac examination:

      * Hereditary long QT syndrome or QTcF>480 msec (the formula is seen in Appendix 10), or currently taking the drugs that are known to prolong QT interval or lead to torsade de pointe arrhythmia (Appendix 6);
      * Serious arrhythmia or conduction abnormality requiring clinical intervention;
      * Impaired cardiac function or clinically significant cardiac disease, including but not limited to the acute myocardial infarction, unstable angina pectoris, coronary artery bypass grafting, New York Heart Association (NYHA, see Appendix 9) evaluated Grade III/IV congestive heart failure, left ventricular ejection fraction (LVEF) <50%, or uncontrollable hypertension within 6 months prior to enrollment.
  11. Pregnant or lactating women;
  12. Having multiple factors affecting absorption, distribution, metabolism or excretion of oral drugs, e.g., inability to swallow, frequent vomiting, chronic diarrhea, etc.;
  13. Currently known or previous retinopathy;
  14. Any other disease, metabolic abnormality, physical examination abnormality or clinically significant laboratory examination abnormality, one disease or state that may affect patient's compliance or provides a reason to suspect that the patient is not suitable to use the study drug, or will affect interpretation of the study results, or bring the patient at a high risk, according to investigator's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of oral HMPL-295S1 monotherapy for patients with advanced solid tumors; | from Cycle 0Day1 up to Cycle1Day28 (each cycle is 28 days)
  Occurrence of Dose Limiting Toxicities (DLTs) During the DLT Observation Period.
Maximum tolerated dose (MTD)of oral HMPL-295S1. | MTD from 1st patient's Cycle 0Day1 (each cycle is 28 days) up to last patient's Last dose in escalation stage. (up to a maximum of approximately 2 years )
  1. Occurrence of Adverse Events (AEs) and Treatment-Related AEs.
  2. Number of Participants With Clinical Significant Changes in Vital Signs, Laboratory Parameters and 12-Lead Electrocardiogram (ECG) Findings.
  3. Incidence of AEs leading to dose interruption, reduction or permanent discontinuation.
Recommended phase II clinical study dose (RP2D) of oral HMPL-295S1. | Baseline up to last patient's last tumor assessment completed in escalation stage. (up to a maximum of approximately 2 years )
  The investigator and the sponsor will determine RP2D jointly based on the following factors:
  1. MTD (if reached)
  2. PK/pharmacokinetics and relevant efficacy and safety.

SECONDARY OUTCOMES:
To investigate the pharmacokinetic (PK) profile of oral HMPL-295S1. | from pre-dose to day 5 of cycle 0. (cycle 0 contains 5 days)
  Plasma peak concentration of HMPL-295S1 (Cmax)
AUCinf (Cycle 0 ) of HMPL-295S1. | from pre-dose to day 5 of cycle 0. (cycle 0 contains 5 days)
  AUCinf: area under the concentration vs. time curve from zero to infinity after single (first)dose.
AUC(0-tlast) (Cycle 0 ) of HMPL-295S1. | from pre-dose to day 5 of cycle 0. (cycle 0 contains 5 days)
  AUC from time zero to the last data point.
Objective Response Rate (ORR) | From baseline to final assessment at end of safety follow-up visit (up to a maximum of approximately 3 years)
  Percentage of patients with Complete Response(CR) or Partial Response(PR) as the best response evaluated in accordance with RECIST 1.1;
Time to response (TTR) | From baseline to final assessment at end of safety follow-up visit (up to a maximum of approximately 3 years)
  the time from the first dose of HMPL-295S1 to the first objective response.
Duration of response (DoR) | From baseline to final assessment at end of safety follow-up visit (up to a maximum of approximately 3 years)
  as the time from the first appearance of CR or PR to PD or death for any reason (whichever comes first), in the patients with objective response;
Disease control rate (DCR) | From baseline to final assessment at end of safety follow-up visit (up to a maximum of approximately 3 years)
  the proportion of patients with CR or PR or stable disease (SD) as the best response, and the duration of SD needs to be ≥6 weeks;
Progression-free survival (PFS) | From baseline to final assessment at end of safety follow-up visit (up to a maximum of approximately 3 years)
  time from the first dose of study treatment to PD or death for any reason, whichever comes first;
Overall survival (OS) | From baseline to final assessment at end of safety follow-up visit (up to a maximum of approximately 3 years)
  time from the first dose of study treatment to death for any reason.

OTHER OUTCOMES:
Exploratory objective: To investigate the pharmacodynamic biomarkers of HMPL-295S1. | pre-dose to 4 hour after dose in Cycle1Day22(each cycle is 28 days)
  Biomarkers in the blood specimen before and after treatment, phosphorylation level of ERK downstream signal ribosome S6 kinase (RSK).

CONTACTS AND LOCATIONS:
Overall Officials: Bin Yang, Study Director — Hutchison Medipharma Limited
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No